CLINICAL TRIAL: NCT05633992
Title: A Phase 3, Randomized, Double-blind, Active Comparator-controlled Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 in Pneumococcal Vaccine-naïve Japanese Adults 65 Years of Age or Older
Brief Title: Safety and Immunogenicity of V116 in Vaccine-naïve Japanese Older Adults (V116-009, STRIDE-9)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V116-009; jRCT2031220551 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- V116 (Experimental): Participants receive a single intramuscular (IM) injection of V116 on Day 1.
  Interventions: Biological: V116
- PPSV23 (Active Comparator): Participants receive a single IM injection of PPSV23 on Day 1.
  Interventions: Biological: PPSV23

INTERVENTIONS:
Biological: V116 — Sterile 0.5 mL solution in prefilled syringe containing 4 μg of each pneumococcal polysaccharide (PnPs) antigen 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 15A, 15C, 16F, 17F, 19A, 20A, 22F, 23A, 23B, 24F, 31, 33F, and 35B.
  Other Names: Pneumococcal 21-valent Conjugate Vaccine
  Arms: V116
Biological: PPSV23 — Sterile 0.5 mL solution in prefilled syringe containing 25 μg of each PnPs antigen 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F.
  Other Names: PNEUMOVAX™23
  Arms: PPSV23

SUMMARY:
This is a phase 3, randomized, double-blind, active comparator-controlled study of the safety, tolerability, and immunogenicity of V116 in pneumococcal vaccine-naïve Japanese adults 65 years of age and older. The polyvalent (23-valent) pneumococcal vaccine, PPSV23, is the active comparator. In addition to studying safety/tolerability, it is hypothesized that, at 30 days postvaccination, the immunogenicity of V116 is noninferior to PPSV23 for the 12 common serotypes in V116 and PPSV23 and the cross-reactive serotype 15B in V116, and that the immunogenicity of V116 is superior to PPSV23 for the unique serotype 15C in V116. It is also hypothesized that V116 is superior to PPSV23 in the percentage of participants with ≥4-fold rise from baseline in the 8 unique V116 serotypes (except for 15C), as measured by serotype-specific opsonophagocytic activity (OPA) geometric mean titers (GMTs).

ELIGIBILITY:
Inclusion Criteria:

* Is Japanese
* For females, is not pregnant or breastfeeding and is either not a participant of childbearing potential (POCBP) or is a POCBP and uses acceptable contraception/abstinence; has a negative highly sensitive pregnancy test (urine or serum) within 24 (urine) or 72 (serum) hours before the first dose of study intervention; and has medical, menstrual, and recent sexual activity history reviewed by the investigator to decrease the chance of inclusion of an early undetected pregnancy

Exclusion Criteria:

* Has a history of invasive pneumococcal disease (IPD) [positive blood culture, positive cerebrospinal fluid culture, or positive culture at another sterile site] or known history of other culture-positive pneumococcal disease within 3 years of Visit 1 (Day 1)
* Has a known hypersensitivity to any component of V116 or PPSV23, including diphtheria toxoid
* Has a known or suspected impairment of immunological function including, but not limited to, a history of congenital or acquired immunodeficiency, documented human immunodeficiency virus (HIV) infection, functional or anatomic asplenia, or history of autoimmune disease
* Has a coagulation disorder contraindicating IM vaccination
* Had a recent febrile illness (defined as oral or tympanic temperature ≥100.4°F [≥38.0°C] or axillary or temporal temperature ≥99.4°F [≥37.4°C]) or received antibiotic therapy for any acute illness occurring <72 hours before receipt of study vaccine
* Has a known malignancy that is progressing or has required active treatment <3 years before enrollment
* Received prior pneumococcal vaccine or is expected to receive any pneumococcal vaccine during the study outside the protocol
* Received systemic corticosteroids (prednisone equivalent of ≥20 mg/day) for ≥14 consecutive days and has not completed intervention ≥14 days before receipt of study vaccine
* Is currently receiving immunosuppressive therapy, including chemotherapeutic agents or other immunotherapies/immunomodulators used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease
* Received any nonlive vaccine ≤14 days before receipt of study vaccine or is scheduled to receive any nonlive vaccine ≤30 days after receipt of study vaccine (inactivated influenza and SARS-CoV2 vaccines may be acceptable)
* Received any live virus vaccine ≤30 days before receipt of study vaccine or is scheduled to receive any live virus vaccine ≤30 days after receipt of study vaccine
* Received a blood transfusion or blood products, including immunoglobulin ≤6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product until the Day 30 postvaccination blood draw is complete

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 450 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (8):
- Japan (8):
  - Medical Corporation Heishinkai OPHAC Hospital ( Site 1008), Osaka, Osaka
  - Medical Corporation Heishinkai OCROM Clinic ( Site 1003), Suita-shi, Osaka
  - P-One Clinic ( Site 1001), Hachiōji, Tokyo
  - Heishinkai Medical Group ToCROM Clinic ( Site 1004), Shinjuku-ku, Tokyo
  - Medical Corporation Shinanokai Shinanozaka Clinic ( Site 1006), Shinjuku-ku, Tokyo
  - Medical Corporation Houeikai Sekino Clinical Pharmacology Clinic ( Site 1005), Toshima City, Tokyo
  - PS Clinic ( Site 1002), Fukuoka
  - Nishikumamoto Hospital ( Site 1007), Kumamoto

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Kishino H, Inoue S, Matsuoka O, Yagi M, Igarashi R, Oshima N, Sawata M, Platt HL. A phase 3 randomized trial (STRIDE-9) to evaluate the safety, tolerability, and immunogenicity of V116, a population-specific pneumococcal conjugate vaccine, in pneumococcal vaccine-naive Japanese adults >/=65 years of age. Vaccine. 2025 Aug 30;62:127456. doi: 10.1016/j.vaccine.2025.127456. Epub 2025 Aug 5. PMID 40763490
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | V116 | PPSV23
Started | 225 | 225
Completed | 225 | 225
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V116 | PPSV23 | Total
Number analyzed (Participants) | 225 | 225 | 450
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (5.7) | 70.9 (5.6) | 70.9 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 96 | 195
  Male | 126 | 129 | 255
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 225 | 225 | 450
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 225 | 225 | 450
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) [Geometric Mean (Full Range); unit: Titers] — OPA GMT for each serotype in V116, estimated using a constrained longitudinal data analysis (cLDA) model. Population: The analysis population consists of all randomized participants who had available baseline data.
  Titers
    Serotype 6A: number analyzed (Participants) | 192 | 205 | 397
    Serotype 6A | 108.5 [19.5 to 3133] | 149.1 [19.5 to 9061] | 127.9 [19.5 to 9061]
    Serotype 15A: number analyzed (Participants) | 194 | 191 | 385
    Serotype 15A | 387.0 [21.0 to 9904] | 416.4 [21.0 to 9477] | 401.3 [21.0 to 9904]
    Serotype 16F: number analyzed (Participants) | 205 | 215 | 420
    Serotype 16F | 820.5 [78.0 to 25880] | 757.9 [78.0 to 25880] | 787.8 [78.0 to 175891]
    Serotype 23A: number analyzed (Participants) | 162 | 152 | 314
    Serotype 23A | 324.0 [21.0 to 14131] | 344.8 [21.0 to 7126] | 333.9 [21.0 to 14131]
    Serotype 23B: number analyzed (Participants) | 207 | 216 | 423
    Serotype 23B | 36.6 [5.0 to 4303] | 41.2 [5.0 to 4834] | 38.9 [5.0 to 4834]
    Serotype 24F: number analyzed (Participants) | 202 | 199 | 401
    Serotype 24F | 627.6 [10.5 to 10682] | 641.9 [10.5 to 8032] | 634.6 [10.5 to 10682]
    Serotype 31: number analyzed (Participants) | 219 | 221 | 440
    Serotype 31 | 129.0 [8.0 to 3765] | 176.5 [8.0 to 71474] | 151.0 [8.0 to 71474]
    Serotype 35B: number analyzed (Participants) | 222 | 221 | 443
    Serotype 35B | 852.6 [12.0 to 12052] | 937.0 [12.0 to 11378] | 893.7 [12.0 to 12052]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-site Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The solicited injection-site AEs assessed were redness/erythema, swelling, and tenderness/pain.
Time Frame: Up to 5 days postvaccination
Population: The analysis population includes all participants who received ≥1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | V116 | PPSV23
Number analyzed (Participants) | 225 | 225
Percentage of participants | 32.9 | 39.1

2. Primary Outcome: Percentage of Participants With Solicited Systemic AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The solicited systemic AEs were muscle pain/myalgia, headache, and tiredness/fatigue.
Time Frame: Up to 5 days postvaccination
Population: The analysis population includes all participants who received ≥1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | V116 | PPSV23
Number analyzed (Participants) | 225 | 225
Percentage of participants | 17.3 | 16.4

3. Primary Outcome: Percentage of Participants With Vaccine-related Serious AEs (SAEs)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is another important medical event. SAEs that were reported to be at least possibly related by the investigator to study vaccination were summarized.
Time Frame: Up to 30 days postvaccination
Population: The analysis population includes all participants who received ≥1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | V116 | PPSV23
Number analyzed (Participants) | 225 | 225
Percentage of participants | 0.0 | 0.0

4. Primary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs)
Description: The serotype-specific OPA GMTs for the 12 common serotypes contained in V116 and PPSV23, the unique serotype 15C in V116, and the cross-reactive serotype 15B were determined using the multiplex opsonophagocytic assay (MOPA).
Time Frame: Day 30 postvaccination
Population: The analysis population consists of all randomized participants without deviations from the protocol that may substantially affect this outcome measure's results.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V116 | PPSV23
Number analyzed (Participants) | 225 | 225
Titers
  Day 30, Serotype 3: number analyzed (Participants) | 206 | 205
  Day 30, Serotype 3 | 155.1 [133.6 to 180.1] | 170.8 [143.9 to 202.9]
  Day 30, Serotype 7F: number analyzed (Participants) | 225 | 224
  Day 30, Serotype 7F | 2675.1 [2312.9 to 3094.0] | 2411.4 [2054.5 to 2830.2]
  Day 30, Serotype 8: number analyzed (Participants) | 223 | 219
  Day 30, Serotype 8 | 1293.3 [1133.8 to 1475.2] | 1142.4 [988.3 to 1320.4]
  Day 30, Serotype 9N: number analyzed (Participants) | 190 | 198
  Day 30, Serotype 9N | 2844.8 [2492.7 to 3246.6] | 2710.5 [2297.6 to 3197.6]
  Day 30, Serotype 10A: number analyzed (Participants) | 218 | 216
  Day 30, Serotype 10A | 1591.2 [1367.4 to 1851.7] | 880.2 [690.1 to 1122.6]
  Day 30, Serotype 11A: number analyzed (Participants) | 218 | 214
  Day 30, Serotype 11A | 1269.6 [1057.6 to 1524.1] | 887.9 [748.3 to 1053.4]
  Day 30, Serotype 12F: number analyzed (Participants) | 222 | 216
  Day 30, Serotype 12F | 968.5 [792.5 to 1183.6] | 503.7 [383.8 to 661.0]
  Day 30, Serotype 17F: number analyzed (Participants) | 203 | 203
  Day 30, Serotype 17F | 3138.1 [2673.0 to 3684.2] | 1860.3 [1551.8 to 2230.1]
  Day 30, Serotype 19A: number analyzed (Participants) | 225 | 223
  Day 30, Serotype 19A | 1338.4 [1144.3 to 1565.4] | 1140.7 [925.1 to 1406.5]
  Day 30, Serotype 20A: number analyzed (Participants) | 217 | 205
  Day 30, Serotype 20A | 2617.2 [2212.9 to 3095.5] | 1731.5 [1474.1 to 2033.7]
  Day 30, Serotype 22F: number analyzed (Participants) | 222 | 220
  Day 30, Serotype 22F | 1830.9 [1562.4 to 2145.6] | 1295.5 [1072.6 to 1564.8]
  Day 30, Serotype 33F: number analyzed (Participants) | 221 | 217
  Day 30, Serotype 33F | 7692.4 [6349.4 to 9319.4] | 8610.8 [7029.9 to 10547.1]
  Day 30, Serotype 15C: number analyzed (Participants) | 216 | 203
  Day 30, Serotype 15C | 2488.5 [1993.5 to 3106.6] | 1185.0 [954.1 to 1471.7]
  Day 30, Serotype 15B: number analyzed (Participants) | 207 | 210
  Day 30, Serotype 15B | 2081.1 [1675.0 to 2585.7] | 1479.7 [1218.0 to 1797.5]
  Baseline, Serotype 3: number analyzed (Participants) | 205 | 214
  Baseline, Serotype 3 | 14.2 [12.5 to 16.1] | 14.9 [13.1 to 17.0]
  Baseline, Serotype 7F: number analyzed (Participants) | 216 | 218
  Baseline, Serotype 7F | 243.9 [190.8 to 311.7] | 217.6 [168.8 to 280.4]
  Baseline, Serotype 8: number analyzed (Participants) | 215 | 217
  Baseline, Serotype 8 | 48.8 [38.3 to 62.3] | 46.3 [36.7 to 58.5]
  Baseline, Serotype 9N: number analyzed (Participants) | 209 | 201
  Baseline, Serotype 9N | 383.1 [313.3 to 468.4] | 383.2 [314.6 to 466.8]
  Baseline, Serotype 10A: number analyzed (Participants) | 208 | 199
  Baseline, Serotype 10A | 131.5 [101.3 to 170.6] | 103.5 [77.4 to 138.5]
  Baseline, Serotype 11A: number analyzed (Participants) | 208 | 207
  Baseline, Serotype 11A | 75.2 [55.9 to 101.3] | 91.2 [68.3 to 121.7]
  Baseline, Serotype 12F: number analyzed (Participants) | 219 | 214
  Baseline, Serotype 12F | 18.1 [14.7 to 22.3] | 19.2 [15.6 to 23.7]
  Baseline, Serotype 17F: number analyzed (Participants) | 207 | 211
  Baseline, Serotype 17F | 285.8 [225.7 to 361.8] | 226.8 [181.0 to 284.1]
  Baseline, Serotype 19A: number analyzed (Participants) | 217 | 215
  Baseline, Serotype 19A | 188.1 [151.9 to 232.8] | 179.7 [143.4 to 225.1]
  Baseline, Serotype 20A: number analyzed (Participants) | 210 | 215
  Baseline, Serotype 20A | 460.0 [384.4 to 550.6] | 421.1 [348.9 to 508.1]
  Baseline, Serotype 22F: number analyzed (Participants) | 211 | 203
  Baseline, Serotype 22F | 179.9 [138.0 to 234.7] | 167.9 [128.0 to 220.3]
  Baseline, Serotype 33F: number analyzed (Participants) | 216 | 223
  Baseline, Serotype 33F | 1236.7 [1048.1 to 1459.3] | 1198.9 [1004.3 to 1431.3]
  Baseline, Serotype 15C: number analyzed (Participants) | 207 | 212
  Baseline, Serotype 15C | 110.0 [85.2 to 142.1] | 102.6 [79.4 to 132.4]
  Baseline, Serotype 15B: number analyzed (Participants) | 203 | 196
  Baseline, Serotype 15B | 243.3 [194.6 to 304.1] | 251.7 [199.7 to 317.2]
Statistical Analysis 1: Comparison: V116 vs PPSV23; Serotype 3; Test type: Non-Inferiority — For the 12 serotypes common to both V116 and PPSV23, a conclusion of non-inferiority of V116 to PPSV23 requires the lower bound of the 2-sided 95% confidence interval of the OPA GMT ratio (V116/PPSV23) to be >0.5 (one-sided p-value <0.025); p < 0.001, Constrained Longitudinal Data Analysis; cLDA model with terms for vaccination group, time, interaction of time-by-vaccination, age stratum at baseline, and interaction of time-by-age stratum; Day 30 GMT Ratio = 0.94, 95% CI 2-sided [0.75 to 1.17] — Ratio is V116/PPSV23. GMT ratio and confidence interval estimated from the cLDA model. The cLDA model-based ratio includes estimated data for participants who had baseline data available but no day 30 measurement
Statistical Analysis 2: Comparison: V116 vs PPSV23; Serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 1.08, 95% CI 2-sided [0.88 to 1.33] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: V116 vs PPSV23; Serotype 8; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 1.12, 95% CI 2-sided [0.93 to 1.36] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: V116 vs PPSV23; Serotype 9N; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 1.05, 95% CI 2-sided [0.86 to 1.29] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: V116 vs PPSV23; Serotype 10A; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 1.65, 95% CI 2-sided [1.28 to 2.14] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: V116 vs PPSV23; Serotype 11A; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 1.52, 95% CI 2-sided [1.20 to 1.92] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: V116 vs PPSV23; Serotype 12F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 1.97, 95% CI 2-sided [1.43 to 2.72] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: V116 vs PPSV23; Serotype 17F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 1.60, 95% CI 2-sided [1.28 to 2.00] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: V116 vs PPSV23; Serotype 19A; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 1.16, 95% CI 2-sided [0.93 to 1.45] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: V116 vs PPSV23; Serotype 20A; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 1.44, 95% CI 2-sided [1.18 to 1.77] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 11: Comparison: V116 vs PPSV23; Serotype 22F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 1.39, 95% CI 2-sided [1.10 to 1.76] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 12: Comparison: V116 vs PPSV23; Serotype 33F; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 0.87, 95% CI 2-sided [0.68 to 1.12] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 13: Comparison: V116 vs PPSV23; Serotype 15B; Test type: Non-Inferiority — For serotype 15B, a conclusion of non-inferiority of V116 to PPSV23 requires the lower bound of the 2-sided 95% confidence interval of the OPA GMT ratio (V116/PPSV23) to be >0.5 (one-sided p-value <0.025); p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 1.43, 95% CI 2-sided [1.07 to 1.89] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 14: Comparison: V116 vs PPSV23; Serotype 15C; Test type: Superiority — For serotype 15C, a conclusion of superiority of V116 to PPSV23 requires the lower bound of the 2-sided 95% confidence interval of the OPA GMT ratio (V116/PPSV23) to be >1.0 (one-sided p-value <0.025); p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 4, analysis 1]; Day 30 GMT Ratio = 2.05, 95% CI 2-sided [1.56 to 2.70] — [estimate comment as in outcome 4, analysis 1]

5. Primary Outcome: Percentage of Participants With ≥4-fold Rise From Baseline in Serotype-specific OPAs (Unique to V116)
Description: The percentage of participants with ≥4-fold rise from baseline in serotype-specific OPAs for the 8 unique serotypes contained in V116 (except for 15C) were determined.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: The analysis population consists of all randomized participants without deviations from the protocol that may substantially affect this outcome measure's results, and who had data for both time points.
Measure: Number; unit: Percentage of Participants
Arm/Group | V116 | PPSV23
Number analyzed (Participants) | 225 | 224
Percentage of Participants
  Serotype 6A: number analyzed (Participants) | 184 | 190
  Serotype 6A | 72.8 | 45.3
  Serotype 15A: number analyzed (Participants) | 181 | 169
  Serotype 15A | 59.7 | 26.0
  Serotype 16F: number analyzed (Participants) | 197 | 201
  Serotype 16F | 50.3 | 11.9
  Serotype 23A: number analyzed (Participants) | 144 | 111
  Serotype 23A | 57.6 | 27.9
  Serotype 23B: number analyzed (Participants) | 201 | 199
  Serotype 23B | 82.1 | 43.7
  Serotype 24F: number analyzed (Participants) | 198 | 175
  Serotype 24F | 42.9 | 16.0
  Serotype 31: number analyzed (Participants) | 219 | 214
  Serotype 31 | 70.3 | 13.1
  Serotype 35B: number analyzed (Participants) | 221 | 218
  Serotype 35B | 52.9 | 6.0
Statistical Analysis 1: Comparison: V116 vs PPSV23; Serotype 6A; Test type: Superiority — A conclusion of superiority of V116 to PPSV23 requires the lower bound of the 2-sided 95% confidence interval of the difference (V116-PPSV23) between the percentage of participants to be >0 percentage points (one-sided p-value <0.025); p < 0.001, Stratified Miettinen & Nurminen; Difference in Percent = 27.6, 95% CI 2-sided [17.8 to 36.9] — Estimated difference and confidence interval are based on the Miettinen & Nurminen method
Statistical Analysis 2: Comparison: V116 vs PPSV23; Serotype 15A; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen; Difference in Percent = 33.7, 95% CI 2-sided [23.6 to 43.0] — Estimated difference and confidence interval are based on the Miettinen & Nurminen method
Statistical Analysis 3: Comparison: V116 vs PPSV23; Serotype 16F; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen; Difference in Percent = 38.3, 95% CI 2-sided [29.8 to 46.4] — Estimated difference and confidence interval are based on the Miettinen & Nurminen method
Statistical Analysis 4: Comparison: V116 vs PPSV23; Serotype 23A; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen; Difference in Percent = 29.5, 95% CI 2-sided [17.4 to 40.6] — Estimated difference and confidence interval are based on the Miettinen & Nurminen method
Statistical Analysis 5: Comparison: V116 vs PPSV23; Serotype 23B; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen; Difference in Percent = 38.3, 95% CI 2-sided [29.3 to 46.7] — Estimated difference and confidence interval are based on the Miettinen & Nurminen method
Statistical Analysis 6: Comparison: V116 vs PPSV23; Serotype 24F; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen; Difference in Percent = 27.1, 95% CI 2-sided [18.3 to 35.6] — Estimated difference and confidence interval are based on the Miettinen & Nurminen method
Statistical Analysis 7: Comparison: V116 vs PPSV23; Serotype 31; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen; Difference in Percent = 57.3, 95% CI 2-sided [49.3 to 64.4] — Estimated difference and confidence interval are based on the Miettinen & Nurminen method
Statistical Analysis 8: Comparison: V116 vs PPSV23; Serotype 35B; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.001, Stratified Miettinen & Nurminen; Difference in Percent = 47.0, 95% CI 2-sided [39.5 to 54.1] — Estimated difference and confidence interval are based on the Miettinen & Nurminen method

6. Secondary Outcome: Serotype-specific OPA GMTs (Unique Serotypes)
Description: The serotype-specific OPA GMTs for the 8 unique serotypes contained in V116 (except for serotype 15C) and the cross-reactive serotype 6C in V116 were determined using MOPA.
Time Frame: Day 30 postvaccination
Population: The analysis population consists of all randomized participants without deviations from the protocol that may substantially affect this outcome measure's results, and who had data available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V116 | PPSV23
Number analyzed (Participants) | 225 | 224
Titers
  Serotype 6A: number analyzed (Participants) | 215 | 209
  Serotype 6A | 1263.8 [1036.6 to 1540.7] | 641.8 [507.0 to 812.4]
  Serotype 15A: number analyzed (Participants) | 211 | 197
  Serotype 15A | 2752.3 [2319.8 to 3265.5] | 832.2 [687.4 to 1007.6]
  Serotype 16F: number analyzed (Participants) | 217 | 211
  Serotype 16F | 4094.8 [3574.8 to 4690.4] | 1183.9 [987.2 to 1419.7]
  Serotype 23A: number analyzed (Participants) | 200 | 153
  Serotype 23A | 2107.5 [1702.3 to 2609.1] | 729.2 [556.8 to 955.0]
  Serotype 23B: number analyzed (Participants) | 217 | 206
  Serotype 23B | 1359.0 [1086.7 to 1699.5] | 202.2 [146.5 to 279.2]
  Serotype 24F: number analyzed (Participants) | 221 | 194
  Serotype 24F | 2521.9 [2246.2 to 2831.4] | 1043.8 [878.1 to 1240.7]
  Serotype 31: number analyzed (Participants) | 225 | 218
  Serotype 31 | 2095.4 [1746.3 to 2514.2] | 260.7 [200.9 to 338.2]
  Serotype 35B: number analyzed (Participants) | 224 | 222
  Serotype 35B | 4758.1 [4146.5 to 5459.9] | 1051.4 [886.6 to 1246.9]

7. Secondary Outcome: Serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs)
Description: The GMCs for serotype-specific IgG antibodies were determined using pneumococcal electrochemiluminescence (PnECL).
Time Frame: Day 30 postvaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V116 | PPSV23
Number analyzed (Participants) | 225 | 225
µg/mL
  Serotype 3 | 0.54 [0.47 to 0.61] | 0.58 [0.51 to 0.67]
  Serotype 7F | 6.12 [5.13 to 7.31] | 4.25 [3.50 to 5.14]
  Serotype 8 | 8.13 [7.01 to 9.42] | 6.72 [5.87 to 7.71]
  Serotype 9N | 7.49 [6.23 to 9.01] | 5.44 [4.55 to 6.50]
  Serotype 10A | 8.21 [6.64 to 10.15] | 3.84 [3.09 to 4.79]
  Serotype 11A | 6.00 [5.09 to 7.08] | 3.02 [2.59 to 3.52]
  Serotype 12F | 1.55 [1.23 to 1.95] | 0.66 [0.52 to 0.84]
  Serotype 17F | 10.48 [8.77 to 12.52] | 5.08 [4.32 to 5.98]
  Serotype 19A | 5.70 [4.80 to 6.76] | 4.87 [4.07 to 5.83]
  Serotype 20A | 15.61 [13.20 to 18.47] | 9.78 [8.09 to 11.83]
  Serotype 22F | 2.84 [2.28 to 3.52] | 1.39 [1.14 to 1.69]
  Serotype 33F | 13.93 [11.92 to 16.27] | 12.67 [10.90 to 14.74]
  Serotype 6A | 3.42 [2.74 to 4.26] | 1.64 [1.33 to 2.02]
  Serotype 15A | 9.98 [8.14 to 12.25] | 1.64 [1.35 to 1.98]
  Serotype 15C | 9.87 [7.95 to 12.26] | 4.55 [3.69 to 5.60]
  Serotype 16F: number analyzed (Participants) | 225 | 224
  Serotype 16F | 3.07 [2.56 to 3.68] | 0.37 [0.31 to 0.43]
  Serotype 23A | 2.00 [1.60 to 2.51] | 0.32 [0.27 to 0.39]
  Serotype 23B | 4.22 [3.58 to 4.99] | 1.65 [1.37 to 1.98]
  Serotype 24F | 7.79 [6.26 to 9.71] | 0.41 [0.35 to 0.47]
  Serotype 31 | 2.57 [2.16 to 3.07] | 0.40 [0.34 to 0.46]
  Serotype 35B | 14.19 [12.01 to 16.76] | 1.38 [1.19 to 1.60]
  Serotype 6C | 1.19 [0.97 to 1.46] | 0.50 [0.42 to 0.59]
  Serotype 15B | 10.15 [8.35 to 12.35] | 9.86 [8.40 to 11.59]

8. Secondary Outcome: Serotype-specific Geometric Mean Fold Rise (GMFR) in OPA GMT
Description: The GMFR from baseline in serotype-specific OPA GMTs was determined using MOPA. GMFR is defined as the geometric mean of the ratio of concentration at Day 30 after vaccination divided by concentration at baseline.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V116 | PPSV23
Number analyzed (Participants) | 225 | 224
Ratio
  Serotype 3: number analyzed (Participants) | 187 | 195
  Serotype 3 | 7.2 [6.1 to 8.5] | 7.2 [6.1 to 8.5]
  Serotype 7F: number analyzed (Participants) | 216 | 217
  Serotype 7F | 10.0 [8.0 to 12.6] | 9.8 [8.0 to 12.1]
  Serotype 8: number analyzed (Participants) | 213 | 211
  Serotype 8 | 20.6 [16.4 to 25.8] | 19.1 [15.5 to 23.7]
  Serotype 9N: number analyzed (Participants) | 177 | 177
  Serotype 9N | 6.9 [5.6 to 8.5] | 6.6 [5.3 to 8.1]
  Serotype 10A: number analyzed (Participants) | 202 | 191
  Serotype 10A | 10.1 [8.2 to 12.4] | 7.6 [5.9 to 9.9]
  Serotype 11A: number analyzed (Participants) | 202 | 197
  Serotype 11A | 13.6 [10.5 to 17.7] | 7.3 [5.7 to 9.4]
  Serotype 12F: number analyzed (Participants) | 216 | 206
  Serotype 12F | 32.2 [25.7 to 40.3] | 17.1 [13.2 to 22.1]
  Serotype 17F: number analyzed (Participants) | 186 | 190
  Serotype 17F | 9.8 [7.8 to 12.4] | 7.1 [5.9 to 8.6]
  Serotype 19A: number analyzed (Participants) | 217 | 213
  Serotype 19A | 6.7 [5.5 to 8.1] | 5.8 [4.8 to 6.9]
  Serotype 20A: number analyzed (Participants) | 205 | 196
  Serotype 20A | 5.6 [4.7 to 6.6] | 4.1 [3.4 to 4.8]
  Serotype 22F: number analyzed (Participants) | 208 | 199
  Serotype 22F | 8.9 [6.9 to 11.5] | 6.9 [5.4 to 8.8]
  Serotype 33F: number analyzed (Participants) | 212 | 215
  Serotype 33F | 6.4 [5.2 to 7.8] | 7.3 [6.0 to 8.8]
  Serotype 6A: number analyzed (Participants) | 184 | 190
  Serotype 6A | 9.4 [7.5 to 11.6] | 3.7 [3.0 to 4.5]
  Serotype 15A: number analyzed (Participants) | 181 | 169
  Serotype 15A | 6.7 [5.3 to 8.5] | 2.0 [1.6 to 2.4]
  Serotype 15C: number analyzed (Participants) | 200 | 191
  Serotype 15C | 19.1 [15.2 to 24.1] | 9.3 [7.4 to 11.7]
  Serotype 16F: number analyzed (Participants) | 197 | 201
  Serotype 16F | 4.7 [4.0 to 5.6] | 1.5 [1.4 to 1.7]
  Serotype 23A: number analyzed (Participants) | 144 | 111
  Serotype 23A | 5.9 [4.2 to 8.2] | 1.8 [1.4 to 2.4]
  Serotype 23B: number analyzed (Participants) | 201 | 199
  Serotype 23B | 26.2 [20.5 to 33.6] | 4.2 [3.3 to 5.4]
  Serotype 24F: number analyzed (Participants) | 198 | 175
  Serotype 24F | 3.8 [3.1 to 4.6] | 1.5 [1.2 to 1.8]
  Serotype 31: number analyzed (Participants) | 219 | 214
  Serotype 31 | 13.6 [10.6 to 17.3] | 1.4 [1.2 to 1.6]
  Serotype 35B: number analyzed (Participants) | 221 | 218
  Serotype 35B | 5.5 [4.6 to 6.5] | 1.2 [1.0 to 1.3]
  Serotype 6C: number analyzed (Participants) | 202 | 197
  Serotype 6C | 2.9 [2.4 to 3.7] | 2.0 [1.7 to 2.3]
  Serotype 15B: number analyzed (Participants) | 186 | 185
  Serotype 15B | 7.4 [5.7 to 9.5] | 4.8 [3.7 to 6.2]

9. Secondary Outcome: Serotype-specific GMFR in IgG GMCs
Description: The GMFR from baseline in GMCs for serotype-specific IgG antibodies was determined using PnECL. GMFR is defined as the geometric mean of the ratio of concentration at Day 30 after vaccination divided by concentration at baseline.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V116 | PPSV23
Number analyzed (Participants) | 225 | 225
Ratio
  Serotype 3 | 5.0 [4.5 to 5.7] | 5.1 [4.5 to 5.8]
  Serotype 7F | 12.1 [10.2 to 14.3] | 8.3 [7.1 to 9.7]
  Serotype 8 | 11.6 [9.8 to 13.7] | 9.8 [8.4 to 11.3]
  Serotype 9N | 11.8 [9.8 to 14.3] | 9.8 [8.4 to 11.5]
  Serotype 10A | 11.4 [9.7 to 13.4] | 6.4 [5.5 to 7.4]
  Serotype 11A | 8.0 [6.8 to 9.4] | 3.9 [3.5 to 4.4]
  Serotype 12F | 11.9 [9.8 to 14.6] | 6.3 [5.2 to 7.5]
  Serotype 17F | 12.9 [10.9 to 15.2] | 7.0 [6.1 to 8.1]
  Serotype 19A | 5.1 [4.3 to 5.9] | 4.2 [3.7 to 4.9]
  Serotype 20A | 9.5 [8.1 to 11.2] | 6.2 [5.4 to 7.2]
  Serotype 22F | 10.7 [8.9 to 12.9] | 5.7 [4.8 to 6.6]
  Serotype 33F | 8.7 [7.4 to 10.2] | 7.7 [6.6 to 8.9]
  Serotype 6A | 10.4 [8.7 to 12.5] | 4.1 [3.6 to 4.7]
  Serotype 15A | 14.0 [11.8 to 16.5] | 2.7 [2.4 to 3.1]
  Serotype 15C | 14.3 [11.8 to 17.3] | 6.9 [5.9 to 8.1]
  Serotype 16F: number analyzed (Participants) | 225 | 224
  Serotype 16F | 12.8 [11.0 to 14.9] | 1.6 [1.5 to 1.7]
  Serotype 23A | 12.0 [10.1 to 14.4] | 2.0 [1.8 to 2.2]
  Serotype 23B | 8.6 [7.5 to 10.0] | 3.1 [2.8 to 3.5]
  Serotype 24F | 18.0 [15.2 to 21.2] | 1.1 [1.0 to 1.1]
  Serotype 31 | 9.1 [8.0 to 10.5] | 1.5 [1.3 to 1.6]
  Serotype 35B | 12.7 [10.8 to 14.8] | 1.1 [1.0 to 1.1]
  Serotype 6C | 2.7 [2.3 to 3.2] | 1.3 [1.2 to 1.4]
  Serotype 15B | 6.8 [5.7 to 8.2] | 7.3 [6.3 to 8.6]

10. Secondary Outcome: Percentage of Participants With ≥4-fold Rise From Baseline in Serotype-specific OPA GMTs (All Serotypes)
Description: Activity for the serotypes contained in V116 and PPSV23 were determined using MOPA. The percentage of participants who had ≥4-fold rise in OPA titers were calculated from baseline to postvaccination.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 | PPSV23
Number analyzed (Participants) | 225 | 224
Percentage of Participants
  Serotype 3: number analyzed (Participants) | 187 | 195
  Serotype 3 | 73.8 [66.9 to 79.9] | 71.3 [64.4 to 77.5]
  Serotype 7F: number analyzed (Participants) | 216 | 217
  Serotype 7F | 68.5 [61.9 to 74.7] | 69.6 [63.0 to 75.6]
  Serotype 8: number analyzed (Participants) | 213 | 211
  Serotype 8 | 79.8 [73.8 to 85.0] | 81.0 [75.1 to 86.1]
  Serotype 9N: number analyzed (Participants) | 177 | 177
  Serotype 9N | 57.6 [50.0 to 65.0] | 58.8 [51.1 to 66.1]
  Serotype 10A: number analyzed (Participants) | 202 | 191
  Serotype 10A | 69.3 [62.4 to 75.6] | 59.7 [52.4 to 66.7]
  Serotype 11A: number analyzed (Participants) | 202 | 197
  Serotype 11A | 69.3 [62.4 to 75.6] | 55.8 [48.6 to 62.9]
  Serotype 12F: number analyzed (Participants) | 216 | 206
  Serotype 12F | 84.3 [78.7 to 88.8] | 74.3 [67.7 to 80.1]
  Serotype 17F: number analyzed (Participants) | 186 | 190
  Serotype 17F | 66.1 [58.8 to 72.9] | 62.6 [55.3 to 69.5]
  Serotype 19A: number analyzed (Participants) | 217 | 213
  Serotype 19A | 58.1 [51.2 to 64.7] | 61.0 [54.1 to 67.6]
  Serotype 20A: number analyzed (Participants) | 205 | 196
  Serotype 20A | 54.1 [47.1 to 61.1] | 42.3 [35.3 to 49.6]
  Serotype 22F: number analyzed (Participants) | 208 | 199
  Serotype 22F | 62.0 [55.0 to 68.6] | 52.3 [45.1 to 59.4]
  Serotype 33F: number analyzed (Participants) | 212 | 215
  Serotype 33F | 58.0 [51.1 to 64.7] | 63.7 [56.9 to 70.2]
  Serotype 6A: number analyzed (Participants) | 184 | 190
  Serotype 6A | 72.8 [65.8 to 79.1] | 45.3 [38.0 to 52.6]
  Serotype 15A: number analyzed (Participants) | 181 | 169
  Serotype 15A | 59.7 [52.1 to 66.9] | 26.0 [19.6 to 33.3]
  Serotype 15C: number analyzed (Participants) | 200 | 191
  Serotype 15C | 81.0 [74.9 to 86.2] | 65.4 [58.2 to 72.2]
  Serotype 16F: number analyzed (Participants) | 197 | 201
  Serotype 16F | 50.3 [43.1 to 57.4] | 11.9 [7.8 to 17.2]
  Serotype 23A: number analyzed (Participants) | 144 | 111
  Serotype 23A | 57.6 [49.1 to 65.8] | 27.9 [19.8 to 37.2]
  Serotype 23B: number analyzed (Participants) | 201 | 199
  Serotype 23B | 82.1 [76.1 to 87.1] | 43.7 [36.7 to 50.9]
  Serotype 24F: number analyzed (Participants) | 198 | 175
  Serotype 24F | 42.9 [35.9 to 50.1] | 16.0 [10.9 to 22.3]
  Serotype 31: number analyzed (Participants) | 219 | 214
  Serotype 31 | 70.3 [63.8 to 76.3] | 13.1 [8.9 to 18.4]
  Serotype 35B: number analyzed (Participants) | 221 | 218
  Serotype 35B | 52.9 [46.1 to 59.7] | 6.0 [3.2 to 10.0]
  Serotype 6C: number analyzed (Participants) | 202 | 197
  Serotype 6C | 34.2 [27.6 to 41.1] | 25.4 [19.5 to 32.1]
  Serotype 15B: number analyzed (Participants) | 186 | 185
  Serotype 15B | 67.2 [60.0 to 73.9] | 54.6 [47.1 to 61.9]

11. Secondary Outcome: Percentage of Participants With ≥4-fold Rise From Baseline in Serotype-specific IgG GMCs (All Serotypes)
Description: Activity for the serotypes contained in V116 and PPSV23 were determined using PnECL. The percentage of participants who had ≥4-fold rise in IgG titers were calculated from baseline to postvaccination.
Time Frame: Baseline (Day 1) and Day 30 postvaccination
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 | PPSV23
Number analyzed (Participants) | 225 | 225
Percentage of Participants
  Serotype 3 | 56.4 [49.7 to 63.0] | 59.6 [52.8 to 66.0]
  Serotype 7F | 77.8 [71.8 to 83.0] | 70.7 [64.2 to 76.5]
  Serotype 8 | 78.7 [72.7 to 83.8] | 78.7 [72.7 to 83.8]
  Serotype 9N | 72.9 [66.6 to 78.6] | 75.1 [68.9 to 80.6]
  Serotype 10A | 79.1 [73.2 to 84.2] | 61.8 [55.1 to 68.2]
  Serotype 11A | 69.3 [62.9 to 75.3] | 44.9 [38.3 to 51.6]
  Serotype 12F | 73.3 [67.0 to 79.0] | 56.9 [50.1 to 63.5]
  Serotype 17F | 82.7 [77.1 to 87.4] | 69.3 [62.9 to 75.3]
  Serotype 19A | 49.3 [42.6 to 56.1] | 47.1 [40.4 to 53.9]
  Serotype 20A | 75.1 [68.9 to 80.6] | 59.6 [52.8 to 66.0]
  Serotype 22F | 71.6 [65.2 to 77.4] | 56.9 [50.1 to 63.5]
  Serotype 33F | 71.6 [65.2 to 77.4] | 73.3 [67.0 to 79.0]
  Serotype 6A | 76.4 [70.3 to 81.8] | 45.8 [39.1 to 52.5]
  Serotype 15A | 80.9 [75.1 to 85.8] | 27.6 [21.8 to 33.9]
  Serotype 15C | 77.8 [71.8 to 83.0] | 61.3 [54.6 to 67.7]
  Serotype 16F: number analyzed (Participants) | 225 | 224
  Serotype 16F | 80.4 [74.7 to 85.4] | 8.0 [4.8 to 12.4]
  Serotype 23A | 76.9 [70.8 to 82.2] | 14.7 [10.3 to 20.0]
  Serotype 23B | 72.9 [66.6 to 78.6] | 35.6 [29.3 to 42.2]
  Serotype 24F | 87.6 [82.5 to 91.6] | 0.0 [0.0 to 1.6]
  Serotype 31 | 75.6 [69.4 to 81.0] | 7.6 [4.5 to 11.8]
  Serotype 35B | 84.0 [78.5 to 88.5] | 0.9 [0.1 to 3.2]
  Serotype 6C | 29.8 [23.9 to 36.2] | 6.7 [3.8 to 10.8]
  Serotype 15B | 60.4 [53.7 to 66.9] | 65.3 [58.7 to 71.5]

ADVERSE EVENTS:
Time Frame: Up to approximately 30 days
Description: All participants who received at least 1 dose of study intervention are included.
Arm/Group | V116 | PPSV23
All-Cause Mortality (participants affected / at risk) | 0/225 | 0/225
Serious Adverse Events (participants affected / at risk) | 1/225 | 0/225
Other Adverse Events (participants affected / at risk) | 77/225 | 96/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V116 (N=225) | PPSV23 (N=225)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V116 (N=225) | PPSV23 (N=225)
Injection site pain (General disorders) | 60 (60) | 81 (82)
Injection site erythema (General disorders) | 19 (19) | 24 (24)
Fatigue (General disorders) | 15 (15) | 25 (25)
Injection site swelling (General disorders) | 14 (14) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT05633992/Prot_SAP_000.pdf